CLINICAL TRIAL: NCT00005820
Title: A Phase II Study of 9 Nitrocamptothecin for Hormone Refractory Prostate Cancer
Brief Title: Nitrocamptothecin in Treating Patients With Stage IV Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-99901; U10CA031946 (NIH); CLB-99901; GUMC-00192; CDR0000067827 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2000-06-02; First posted 2004-04-12 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nitrocamptothecin (Experimental): Patients receive nitrocamptothecin orally daily for 5 consecutive days each week for 3 consecutive weeks. Treatment continues every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 3 months until evidence of progression or relapse for a maximum of 2 years from the date of registration.
  Interventions: Drug: nitrocamptothecin

INTERVENTIONS:
Drug: nitrocamptothecin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of nitrocamptothecin in treating men who have stage IV prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the therapeutic efficacy of nitrocamptothecin in patients with metastatic, hormone refractory prostate cancer.
* Determine time to disease progression and duration of response in this patient population as a result of this treatment regimen.
* Determine the safety, tolerance, and toxicity of this treatment regimen in these patients.

OUTLINE: Patients receive nitrocamptothecin orally daily for 5 consecutive days each week for 3 consecutive weeks. Treatment continues every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months until evidence of progression or relapse for a maximum of 2 years from the date of registration.

PROJECTED ACCRUAL: A total of 22-46 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate with clinically progressive stage IVA or IVB disease after at least primary androgen ablation with either orchiectomy or LHRH agonist and only one cytotoxic chemotherapy regimen
* Measurable disease with a maximum of 10 measurable lesions OR nonmeasurable disease
* Serum testosterone no greater than 50 ng/mL if no prior bilateral orchiectomy

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* ECOG 0 or 1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3 (transfusion independent)
* No disseminated intravascular coagulation

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 3 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* Fertile patients must use effective contraception
* No currently active second malignancy other than nonmelanoma skin cancers
* No active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered

Chemotherapy:

* See Disease Characteristics
* At least 6 weeks since prior suramin
* At least 4 weeks since other prior chemotherapy
* No prior therapy with camptothecin or any of its analogues

Endocrine therapy:

* Prior second line hormonal therapy allowed
* At least 4 weeks since prior hormonal therapy
* Concurrent treatment with LHRH agonists allowed and required for
* patients without orchiectomy
* No concurrent hormonal therapy except for nondisease related conditions
* Concurrent corticosteroids allowed if on stable dose for at least 6 weeks
* before study
* No concurrent dexamethasone as an antiemetic

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered
* No palliative radiotherapy
* At least 8 weeks since prior strontium 89 or samarium 153

Surgery:

* At least 3 weeks since major surgery and recovered

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2000-05; Primary Completion 2004-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
median time to disease and PSA progression | Up to 2 years

SECONDARY OUTCOMES:
overall survival | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Edward P. Gelmann, MD, Study Chair — Lombardi Comprehensive Cancer Center
Locations (50):
- United States (50):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Amin A, Halabi S, Gelmann EP, Stadler W, Vogelzang N, Small E. 9-Nitrocamptothecin as second line chemotherapy for men with progressive, metastatic, hormone refractory prostate cancer: Results of the CALGB 99901. Urol Oncol. 2004 Sep-Oct;22(5):398-403. doi: 10.1016/j.urolonc.2004.05.002. PMID 15464920